CLINICAL TRIAL: NCT04726995
Title: Efficacy and Safety Comparison Between R-CHOP/CHOP and Modified NHL-BFM-90 Regimens in Children and Adolescents With Diffuse Large B-cell Lymphoma
Brief Title: DLBCL Treatment in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhuo Zhang, professor, Sun Yat-sen University
Other Study IDs: DLBCL treatment
Record Dates: First submitted 2021-01-21; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Diffuse Large B-cell Lymphoma
Keywords: Children, Adolescent, Treatment, Modified NHL-BFM-90, R-CHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CHOP and BFM regiments — used CHOP and BFM regiments

SUMMARY:
We compared the efficacy and safety of modified NHL-BFM-90 regimen and R-CHOP/CHOP regimen in pediatric (aged 0-14 years) and adolescent（aged 15-18 years）DLBCL patients in a single institution during a 20-year period. we compared the efficacy and safety of modified NHL-BFM-90 regimen and R-CHOP/CHOP regimen in pediatric (aged 0-14 years) and adolescent（aged 15-18 years）DLBCL patients in a single institution during a 20-year period. To our best knowledge, no reports have been previously published regarding the comparison.

DETAILED DESCRIPTION:
Diffuse large B-cell lymphoma (DLBCL) is an aggressive lymphoma that accounts for approximately 10%-20% of pediatric and adolescent non-Hodgkin's lymphomas (NHLs).

The incidence increases with age, with 37% of NHLs patients being adolescents aged. Poor survival has been demonstrated in adolescents and young adults compared to children with DLBCL. However, the Associazione Italiana Ematologia Oncologia Pediatrica (AIEOP) LNH-97 study showed that age was not a poor prognostic factor in children and adolescents with Burkitt lymphoma (BL) and DLBCL. A conclusion as to whether adolescent age is an independent risk factor has not been reached.

At present, the preferred protocols for adolescent DLBCL patients have not been standardized. Adolescents with cancer have been designated as a vulnerable population, positioned between children and the adult population. Treatment strategies differ between adults and pediatric patients. The pediatric strategy for DLBCL was developed in parallel by the Berlin-Frankfurt-Münster (BFM) and French-American-British/Lymphomes Malins B (FAB/LMB) groups. The combination of rituximab plus Cyclophosphamide, Adriamycin, Vincristine, and Prednisone (R-CHOP) or R-CHOP-like chemotherapy regimens are the standard therapy for the treatment of adult patients with DLBCL. There is currently a lack of studies that have compared the treatment outcomes in adolescent patients with DLBCL who were administered pediatric or adult regimens. Hence, we retrospectively analyzed the clinical characteristics and prognostic factors in DLBCL patients, especially the efficacy and safety of the pediatric regimen (modified NHL-BFM-90) and adult regimen (R-CHOP/CHOP), between pediatric and adolescent DLBCL patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients who were pathologically diagnosed with DLBCL
2. patients under 18 years of age.

Exclusion Criteria:

1. Was administered prior chemotherapy;
2. Patients who could not receive chemotherapy due to severe immunodeficiency or other diseases.
3. Patients with primary central nervous system lymphomas.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: DLBCL patients aged 0-18 year-old
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
OS | through study completion, an average of 58 months
  Overall survival (OS) was calculated from the date of diagnosis to death due to any cause or to the date of the last follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhuo Zhang, Principal Investigator — Sun Yat-sen University CancerCenter

IPD SHARING:
Plan to Share IPD: No